CLINICAL TRIAL: NCT06334679
Title: The Effect of Cold Gel Pack Application on Itching in Burn Patients in the Maturation Stage: A Randomized Controlled Study
Brief Title: The Effect of Cold Gel Pack Application on Itching in Burn Patients in the Maturation Stage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Zeynep Ersöz, PhD Candidate, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: zeynepersoz
Record Dates: First submitted 2024-03-08; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Burns; Pruritus
Keywords: Burn; İtch/Pruritus; Cold Application; Maturation; Cold Gel Pack
MeSH Terms: conditions — Burns; Pruritus

STUDY DESIGN:
Intervention Model Description: It is a prospective interventional type two-group randomized controlled clinical study. Distribution according to the groups and layers to be assigned for each intervention; Group-1 (Experiment) was designed as clinical routine (liquid petroleum jelly) and cold gel pack, and Group-2 (Control) was designed as clinical routine (liquid petroleum jelly).
Who Masked: Outcomes Assessor
Masking Description: When cold application studies in the literature are examined, cold gel packs are placed in a sheath and contacted with the skin of the patients. Therefore, due to the nature of the application method to be used, patients and the researcher will not be considered blind. The evaluator will be considered blind in the analysis of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-1 (Clinical Routine (liquid vaseline) and Cold Gel Pack applied group) (Experimental): Before the first application of the day, the "12-Item Itching Severity Scale" will be applied to evaluate the patient's daily itching. Before each application, itching severity will be evaluated with the Visual Analog Scale (VAS) for Itch at minute 0. Vital signs will be measured and recorded. Cold gel packs placed in a sterile cloth sheath will be placed in full contact with the burn areas and applied for 20 minutes. During the application, the skin will be checked every 30 seconds and 5 minutes, and the application will be interrupted in case of new pain, numbness, redness, pallor, chills, cold sensitivity and skin surface temperature ≤13 degrees Celsius. The temperature of the cold gel packs before and during application will be checked with a Digital Infrared Non-Contact Thermometer. Immediately after the application is completed, a 20-minute VAS for itching will be shown and they will be asked to evaluate the severity of the itching they feel instantly.
  Interventions: Other: Cold Gel Packet Application
- Group-2: Clinical routine (liquid petroleum jelly) applied group (control) (No Intervention): Before the first application of the day, the "12-Item Itching Severity Scale" will be applied to evaluate the patient's daily itching. Before each application, the Visual Analog Scale (VAS) for Itch will be shown at minute 0 and they will be asked to evaluate the severity of itching they feel immediately. Vital signs will be measured and recorded. Liquid petroleum jelly, which is the routine practice of the clinic, will be applied by clinic nurses. Immediately after the application is completed, a 20-minute VAS for itching will be shown and they will be asked to evaluate the severity of itching they feel immediately.

INTERVENTIONS:
Other: Cold Gel Packet Application — Cold gel packs will be placed on the burn areas of the patients in the maturation phase and applied for 20 minutes.
  Arms: Group-1 (Clinical Routine (liquid vaseline) and Cold Gel Pack applied group)

SUMMARY:
Burn is a serious trauma that causes acute damage to the skin and subcutaneous tissues due to the effect of heat, electricity, radiation, physical, and chemical substances. It has been reported that the incidence of itching is high in burn patients during the maturation stage of wound healing. The literature suggests that in managing the symptom of itching, skin hydration support along with cold application methods can also be used. The integrity of the skin, the duration, frequency, characteristics, areas of itching, and identifying conditions that increase or decrease itching are important for managing itching. This study is planned to be conducted with a randomized controlled design to examine the effect of applying cold gel packs to burn areas of burn patients during the maturation stage on itching. This researcher's hypothesis is that burn patients who applied cold gel packs to burn areas during the maturation phase had lower itching severity (frequency, duration, intensity) than those who did not.

DETAILED DESCRIPTION:
Patients will be assigned to one of two groups according to the block randomization list, given a sequence number according to the date and time of admission. In addition to the clinical routine application, cold gel pack application will be applied to the patients in Group 1, and the clinical routine application will continue for those in Group 2. To collect data, the Patient Diagnosis Form developed by the researcher in line with literature information, the Visual Analog Scale for Itching, the Bates-Jensen Wound Assessment Tool and the 12-Item Itching Severity Scale, whose validity and reliability analysis has been conducted, will be used. Calculation of the sample size of the study was made with the G.Power (v3.1.7) computer program. In the study of Joo et al., a total of 26 patient samples were used to represent the universe, assuming that the difference in two independent groups was considered statistically significant according to the itching degree averages of burn patients (α = 0.05 significance level and 95% power). During the research process, it was decided to include a total of 60 individuals in the sample, with 30 patients in Group-1 (Experiment) and 30 patients in Group-2 (Control), taking into account possible losses.

ELIGIBILITY:
Inclusion Criteria:

* Burn percentage is between 15-25% and 1st or 2nd degree burn areas are in the maturation phase (BatesJensen Wound Assessment Tool Scale score=1-13),
* Describing itching in burn wounds in the last 24 hours,
* Over 18 years of age,
* Literate,
* Oriented to person, place and time,
* Having no vision, speech or communication problems,
* Do not have any skin disease other than burns,
* Patients whose vital signs are within physiological limits (Pulse: 60-100/min, Temperature: average 37 degrees Celsius, respiration 12-16/min, Blood Pressure: average 120/80).

Exclusion Criteria:

* Cold sensitivity/allergy,
* Perineum, neck and inner wrist burn areas
* Hypertrophic scar area,
* Burn infection
* Raynaud's disease,
* Use of aspirin, anticoagulants, non-steriod anti-inflammatory drugs,
* Evitamin and vasoactive agent use,
* Peripheral vascular disease,
* Connective tissue disease,
* Diabetic neuropathy,
* Use of a medication that will cause itching,
* Patients participating in another study conducted at the clinic
* Applying medical treatment in addition to the clinical routine due to itching,
* Due to the fact that he was discharged in a shorter period of time than the average hospitalization day, the research process failure to complete,
* Failure to comply with the monitoring process and conditions of the research,
* It was determined as the person wanting to leave the study voluntarily.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Itching severity | The itching severity of the patients was measured with the "12-Item Itching Severity Scale"; Before the first application, it will be evaluated a total of 5 times over 4 days, on the morning of the next day of application.
  The scale consists of 12 questions. Questions 2, 3, 4, 5, 6, 7, 8 and 12 in the scale have two options, "yes" and "no", and the scoring changes as 1 or 0. The frequency of itching in the first question and itchy areas in the 11th question are marked and scored between 1 and 3. The 9th question, which evaluates the frequency of waking up from sleep due to itching, has 4 items and is scored between 0-3. The 10th question, which evaluates the severity of itching, has 5 items and is scored between 1-5. The score obtained from the scale is at least 3 and at most 22, and as the score increases, the level of being affected by itching also increases. Scores obtained as a result of the scale indicate mild itching between "3-6", moderate itching between "7-11" and severe itching between "12-22".
Itching grade | itching grade will be evaluated instantly with the Visual Analog Scale (VAS) 0 minutes before each application and 20 minutes immediately after the application.The scale will be evaluated for 4 days with repeated measurements twice a day before and after
  Visual Analog Scale (VAS).It is stated that Visual Analogue Scale (VAS) can be used to measure the severity of itching. VAS is a numerical and one-dimensional scale and is mostly used to obtain an objective result by evaluating the intensity and severity of itching. The scale is scored between 1-10. VAS is a scale that initially ranges from 0 "I have no itching" to 10 "I have very severe itching", with each interval corresponding to one centimeter and given a numerical value. On the scale, 0 points indicate no itching, 1-3 points indicate mild itching, 4-6 points indicate moderate itching, 7-8 points indicate severe itching, and 9 and above points indicate very severe itching.

CONTACTS AND LOCATIONS:
Locations (1):
- Kartal Dr.Lütfi Kırdar City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Joo SY, Kim JB, Cho YS, Cho YS, Seo CH. Effect of cold pack therapy for management of burn scar pruritus: A pilot study. Burns. 2018 Jun;44(4):1005-1010. doi: 10.1016/j.burns.2018.01.011. Epub 2018 Feb 13. PMID 29422437
- [Result] Stepien K, Reich A. The 12-Item Pruritus Severity Scale - Determining the Severity Bands. Front Med (Lausanne). 2020 Dec 17;7:614005. doi: 10.3389/fmed.2020.614005. eCollection 2020. PMID 33392233
- [Result] Reich A, Bozek A, Janiszewska K, Szepietowski JC. 12-Item Pruritus Severity Scale: Development and Validation of New Itch Severity Questionnaire. Biomed Res Int. 2017;2017:3896423. doi: 10.1155/2017/3896423. Epub 2017 Oct 2. PMID 29098154
- [Result] Stander S, Augustin M, Reich A, Blome C, Ebata T, Phan NQ, Szepietowski JC; International Forum for the Study of Itch Special Interest Group Scoring Itch in Clinical Trials. Pruritus assessment in clinical trials: consensus recommendations from the International Forum for the Study of Itch (IFSI) Special Interest Group Scoring Itch in Clinical Trials. Acta Derm Venereol. 2013 Sep 4;93(5):509-14. doi: 10.2340/00015555-1620. PMID 23624777